CLINICAL TRIAL: NCT05501990
Title: Study on the Accessibility and Feasibility of Intelligent Applet for Health Intervention of Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, lei huang, Research Associate Fellow; PI, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RJODLH-001
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health intervention based on intelligent applet (Experimental): Health interventions using electronic applet, including nutrition, psychology, and patient self-management components.
  Interventions: Behavioral: Health intervention based on intelligent applet

INTERVENTIONS:
Behavioral: Health intervention based on intelligent applet — Patients are jointly managed by a MDT team based on the applet. The supportive intervention based on the applet mainly includes three parts: Nutrition, psychology, and patient management which includes four main parts: Cancer patient education, self-management, patient community, and real-time communication.

SUMMARY:
In the 5G era with the revolutionary improvement of network speed, digital medical care has brought great convenience to health services. There is a lack of mobile medical data on cancer care worldwide. We designed an applet based on mobile intelligent electronic devices with a doctor-patient dual interface for the perioperative management of cancer patients and verified its applicability in the general population. This study aims to specifically improve the applet according to the characteristics of cancer patients, use it to accurately manage and intervene cancer patients, and establish a rapid doctor-patient communication platform, hoping to improve prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date informed consent;
* Commit to abide by the research procedures and cooperate with the implementation of the whole research process ;
* Can adhere to and cooperate with research intervention;
* Tumor patients;
* Patients/family members can use smart phones to access the Internet;
* Patients/family members have sufficient cognitive and reading ability;
* No mental illness;
* No serious visual impairment

Exclusion Criteria:

* Equipped with specific devices (such as cardiac pacemaker);
* Those who do not meet the conditions listed in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the applet by cancer patients as assessed by questionnaire | 3 months
  Investigated by a questionnaire with 33 questions, and compared with other mobile medical methods to explore the accessibility
Acceptability of the applet by medical oncology staff as assessed by questionnaire | 3 months
  The questionnaire includes 22 questions, collecting information on attitude feedback, time input, and training cost of medical staff using the mobile medical applet

SECONDARY OUTCOMES:
Self-reported quality of life as assessed by ED-5Q-5L scale | 3 months
  EQ-5D-5L is a set of standardized scales for measuring health status, including 5 dimensions (1-5 points for each dimension) and a VAS for overall assessment of health status. Developed by the European Society for quality of life, it can provide a simple and universal health measurement method for clinical and economic evaluation.
Psychological status as assessed by the HADS scale | 3 months
  Hospital Anxiety and Depression Scale (HADS): A self screening questionnaire composed of 7 anxiety subscales and 7 depression subscales. The total score of each subscale is between 0 and 21. The higher the total score, the more serious the anxiety or depression.
Symptom distress as assessed by the MD Anderson symptom scale | 3 months
  Symptom distress is assessed with MD Anderson symptom scale, which is composed of 13 symptom severity and 6 symptom interference subscales. It is used to assess the interference of symptoms to patients' daily life. The item scores range from 1 to 10. The higher the average score, the more serious the symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Huang, PhD, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital，Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No